CLINICAL TRIAL: NCT01761825
Title: The Effect of "Funny" Channel Blocker Ivabradine on Patients With Postural Tachycardia Syndrome.
Brief Title: The Effect of Ivabradine on Patients With Postural Tachycardia Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-12-JG-547-CTIL
Record Dates: First submitted 2012-11-17; First posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Postural Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ivabradine (Active Comparator): Ivabradine 10 mg once
  Interventions: Drug: ivabradine
- placebo (Placebo Comparator)

INTERVENTIONS:
Drug: ivabradine
  Arms: Ivabradine

SUMMARY:
The purpose of this study is to determine whether Ivabradine is an effective treatment for postural tachycardia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with POTS by the following criteria:

  1. The presence of characteristic orthostatic symptoms of the POTS for at least six months.
  2. An increase in the heart rate of at least 30 beats per minute (without concomitant significant decrease in blood pressure of more than 20/10 mmHg) within 10 minutes after assuming a standing position (or during tilt test) on at least 3 separate occasions.
  3. No other concomitant diseases that could explain the symptoms of POTS.

     Exclusion Criteria:

  <!-- -->

  1. History of systemic illness capable of affecting of affecting autonomic function (eg, diabetes mellitus, SLE).
  2. History of cardiovascular disease.
  3. History of smoking, drug or alcohol abuse.
  4. Pregnancy, and also uncontrolled thyroid or adrenal disorders.
  5. Using any drug metabolized by cytochrome P450 3A4 enzyme during the last 72 hours.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
the change in heart rate after the administration of Ivabradine | 60 minutes , during the whole trial
the change in blood pressure after the administration of Ivabradine | 60 minutes